CLINICAL TRIAL: NCT05812326
Title: Exploratory Clinical Study of PD-1 Knockout Targeting MUC1 CAR-T Cells (AJMUC1) in the Treatment of MUC1-positive Advanced Breast Cancer
Brief Title: PD-1 Knockout Anti-MUC1 CAR-T Cells in the Treatment of Advanced Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: Guangzhou Anjie Biomedical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2019-KY-001-003
Record Dates: First submitted 2022-10-11; First posted 2023-04-13 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2022-10

CONDITIONS: Advanced Breast Cancer; Breast Neoplasm Malignant Female
Keywords: Breast cancer, solid tumor, CAR-T cells, PD-1 knockout, MUC1
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment with AJMUC1--PD-1 knockout CAR-T cells (Experimental): Advanced breast cancer patients with positive MUC1 expression are the indications of this clinical study. Current conventional treatments are ineffective for these patients or there is no effective treatment plan available for them. No control group is established and a single arm design is used.
  This clinical study is the first application of AJMUC1 in the clinical treatment of MUC1-positive advanced breast cancer patients. The main purpose is to assess the safety and feasibility of the product in clinical use. Therefore, according to the principle of "3+3" dose escalation design, this study explored the maximum tolerated dose of AJMUC1 for the treatment of MUC1-positive advanced breast cancer.
  At the same time, the efficacy of AJMUC1 in the treatment of MUC1-positive advanced breast cancer will be observed and factors that could affect the safety and efficacy of the therapy will be exploringly evaluated.
  Interventions: Drug: AJMUC1- PD-1 gene knockout anti-MUC1 CAR-T cells

INTERVENTIONS:
Drug: AJMUC1- PD-1 gene knockout anti-MUC1 CAR-T cells — AJMUC1 is a genetically modified T cell therapeutic product targeting the aberrantly glycosylated MUC1 protein. CAR targeting MUC1 is introduced into autologous T cells by lentiviral vector, so that T cells expressing the receptor can recognize and kill MUC1 positive tumor cells. Preclinical studies have shown that binding of scFv targeting MUC1 to the MUC1 epitope on the surface of the target cell can induce the costimulatory CD28 and CD3ζ costimulatory domains to activate downstream signaling pathways and promote T cell activation and expansion. Activated CAR-T cells secrete a series of inflammatory cytokines and chemokines, leading to apoptosis and necrosis of target tumor cells. Following introduction of a CAR structure, the PD-1 gene of CAR-T cells is knocked out using CRISPR/Cas9, so that the CAR-T cell does not express PD-1, resulting in improved tumor killing efficiency of AJMUC due to the release of inhibition in the signaling pathway PD-1/PD-L1 in the tumor microenvironment.
  Other Names: Therapeutic T cells

SUMMARY:
This exploratory clinical study aims to assess the safety and preliminary efficacy of an immunotherapy using PD-1 knockout anti-MUC1 CAR-T cells in the treatment of advanced MUC1-positive breast cancer

DETAILED DESCRIPTION:
This is a single-center, open-label, dose-escalation exploratory study investigating the safety,tolerability and preliminary efficacy of AJMUC1, PD-1 knockout CAR-T cells targeting aberrantly glycosylated MUC1, in the treatment of patients with advanced MUC1 positive breast cancer. The primary objective of this study is to evaluate the safety, tolerability, biological activity, and preliminary antitumor efficacy of AJMUC1. The study adopts a "3+3" dose escalation design to identify the maximum tolerated dose (MTD)/ maximum administered dose (MAD). Three doses are set: 3×105 CAR T cells/kg, 1×106 CAR T cells/kg and 3×106 CAR T cells/kg, with a total of 15 patients planned by the data cutoff date. Participants may receive one, two, three or more cycles of AJMUC1 infusion dependent on the adverse effects and potential clinical benefits.. This study is initiated by the investigators and approved by the Human Ethics Committee of Sun Yat-sen Memorial Hospital affiliated with Sun Yat-sen University. All patients have signed informed consent.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age: 18-70 years (including the boundary value);
2. Pathologically diagnosed with recurrent/metastatic breast cancer (except for intracranial metastasis), who have received at least one standard treatment regimen in the past, the disease is in a stable or progressive state, and refuses to undergo subsequent chemotherapy;
3. Abnormal glycosylated MUC1 expression confirmed by immunohistochemistry in tumor tissue or puncture tissue within 12 months;
4. Expected survival period ≥ 4 months;
5. ECOG score≤2 points;
6. The subjects voluntarily joined the study, signed the informed consent form, had good compliance, and cooperated with the follow-up;
7. Able to cooperate with tumor puncture;
8. At least one measurable lesion that meets the RECIST v1.1 criteria;
9. Female patients of childbearing age must not be breastfeeding, and serum or urine HCG test is negative within 72 hours before study enrollment. All subjects must use medically approved contraception during the study period and within 3 months after the end of the study. measures (eg, IUDs, birth control pills) for contraception;
10. Organ function and bone marrow reserve are in good condition and the following requirements must be met: (1) The absolute value of neutrophils is ≥1.5×109/L; (2) Platelet count ≥75×109/L; (3) Hemoglobin ≥9g/dl; (4) Bilirubin value < 1.5 times the upper limit of normal (except for obstruction of the bile duct caused by tumor compression); (5) Creatinine value < 1.5 times the upper limit of normal or creatinine clearance rate ≥ 60ml/min; (6) ALT or AST < 2.5 times the upper limit of normal (with liver involvement < 5 times the upper limit of normal); (7) Stable coagulation function: INR≤1.5, PTT<1.2 times the upper limit of normal (except for tumor-related anticoagulation therapy).

Exclusion Criteria:

1. Have used immunosuppressive drugs or hormones within 1 week prior to enrollment;
2. Patients with moderate or more moderate pleural and ascites who need catheter drainage to relieve symptoms;
3. Human immunodeficiency virus (HIV) positive;
4. Active hepatitis B or C infection;
5. Pregnant or lactating women;
6. Past or concurrent history of other malignant tumors. Excluded: Patients with basal or squamous cell carcinoma of the skin and carcinoma in situ of the cervix who have been cured at any time prior to the study;
7. Those with central transfer;
8. Serious, uncontrollable concomitant diseases that may affect protocol compliance or interfere with the interpretation of results, or have any serious medical conditions that may affect the subject's safety (such as uncontrollable heart disease, high blood pressure, active or uncontrollable disease) infection, etc.);
9. Active autoimmune diseases (including but not limited to, systemic lupus erythematosus, Sjögren syndrome, rheumatoid arthritis, psoriasis, multiple sclerosis, inflammatory bowel disease, etc.);
10. Those with a history of organ transplantation;
11. Subjects whose last medication was less than 2 weeks before enrollment, or subjects who participated in other relevant clinical studies at the same time;
12. Those who have received gene therapy in the past;
13. Vaccination with live vaccine within 4 weeks prior to study;
14. History of myocardial infarction and severe arrhythmia within half a year; uncontrolled hypertension, coronary heart disease, stroke, liver cirrhosis, nephritis and other serious complications;
15. Those who have a history of psychotropic substance abuse and cannot quit or who have a history of mental disorders;
16. Hypersensitivity constitution, allergic to human serum albumin;
17. Hemorrhagic and thrombotic tendency: patients with clinically significant bleeding symptoms or clear bleeding tendency within 3 months before the study, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, abnormal coagulation function (PT>16s, APTT>43s) , TT>21s, FIB<2g/L), hereditary or acquired bleeding and thrombosis tendency to (such as hemophilia, coagulation disorder, thrombocytopenia, hypersplenism, etc.), are receiving thrombolytic or anticoagulation therapy, arterial/venous thrombotic events occurred within the previous 6 months, such as cerebrovascular disease (including cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism;
18. Other severe, acute, or chronic medical or psychiatric conditions that may increase the risks associated with participation in the study or may interfere with the interpretation of the study results, in the opinion of the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-05-17 (Actual); Primary Completion 2022-11-16 (Actual); Study Completion 2022-11-16 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events and dose limiting toxicities as assessed by CTCAE v5.0 | 3 years
Incidence of treatment-emergent adverse events [safety and tolerability] of dose of PD-1 Knockout CAR-T cells will be assessed using CTCAE v5.0 | 3 years
Monitoring the numbers of circulating AJMUC1 after infusion will be evaluated. | up to 3 years

SECONDARY OUTCOMES:
Response rate will be assessed according to the revised RECIST guideline iRECIST | 3 years
Overall Survival - OS (Measure the time from enrollment to death) | 3 years
Progression free survival - PFS (Time from enrollment to date of first documented progression or date of death) | 3 years
Median CAR-T cell persistence--Will be measured by quantitative RT-PCR | 3 years

OTHER OUTCOMES:
To evaluate serum cytokine changes after AJMUC1 treatment of aberrantly glycosylated MUC1 expression in advanced breast cancer | 3 years
  The serum cytokine included IL-1β, IL-2R, IL-6, IL-8, TNF and IL-10

CONTACTS AND LOCATIONS:
Overall Officials: Erwei Song, MD, PhD, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Hospital Website--Sun Yat-sen Memorial Hospital of Sun Yat-sen University — http://www.gzsys.org.cn/en/home
- See also: Company Producing CAR-T Cell Products--Guangzhou Anjie Biomedical Technology Co. Ltd — http://www.anjiebiomed.com/